CLINICAL TRIAL: NCT06041412
Title: The Effect of Related Blood Markers on Diabetic Peripheral Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: DPN
Record Dates: First submitted 2022-12-26; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Peripheral Neuropathy; electromyography; blood parameters

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DPN group: Patients with type 2 diabetic peripheral neuropathy were categorized into the DPN group
- Diabetic group: patients with type 2 diabetes mellitus but not with DPN were distributed into the Diabetic group.
- control group: The other individuals without type 2 diabetes mellitus were selected as the control group

SUMMARY:
The goal of this observational study is to explore the relationship between related blood indicators and diabetic peripheral neuropathy(DPN).

DETAILED DESCRIPTION:
This is a multicenter study(approximately four) with over 1000 subjects.Clinical data were collected by consulting the patient's electronic history. The data included demographic information, blood biochemical markers and electromyography. All participants provided their written informed consent to participate in this study.The study protocol was approved by the Ethics Committee of the First Affiliated Hospital of Wenzhou Medical University(KY-2022-R009).

ELIGIBILITY:
Inclusion Criteria:

* patients who had undergone nerve conduction examination by electromyography.

Exclusion Criteria:

* pregnancy and lactation; chronic liver disease, kidney disease, arrhythmias, malignant diseases, severe respiratory diseases, heart failure, and acute infections;
* patients with alcohol abuse; history of Autoimmune liver disease, liver disease or abnormal liver function at baseline;
* parathyroid diseases (including hyperthyroidism and hypothyroidism);
* pancreatitis, pancreatectomy or any transplant;
* patients with malignancy and any serious concomitant disease limit the existence of life expectancy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a multicenter study(approximately four) with over 1000 subjects.Clinical data were collected by consulting the patient's electronic history. The data included demographic information, blood biochemical markers and electromyography. All participants provided their written informed consent to participate in this study.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
the severity of DPN | From admission to discharge, up to 1 week
  The nerve conduction examination was conducted at a room temperature of 24℃, with the legs warmed using an electric heating pad for at least 10 minutes to achieve a skin temperature of 32-35℃. The nerve conduction velocities and nerve conduction amplitudes were measured for both sides of the upper and lower limbs, including motor and sensory branches of the median nerve; motor and sensory branches of the ulnar nerve; motor branch of peroneal nerve; motor branch of the tibial nerve; sensory branch of the superficial peroneal nerve. In addition, both sides of the tibial nerve F-wave were recorded, and the lower one was regarded as the final F-wave. Slowed/blocked nerve conduction was defined as more than 2.5 standard deviation below the control nerve conduction threshold. Nerve conduction is defined as abnormal when two or more nerve abnormalities are detected.
the presence of DPN | From admission to discharge, up to 1 week
  When any of the elements of the screening process -- symptoms, signs, or abnormal nerve conduction parameters --was abnormal, medical records would be scrutinized to see if these participants had accepted a previous DPN diagnosis by a specialist.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China